CLINICAL TRIAL: NCT03784781
Title: Type 2 Innate Lymphoid Cells in Severe Pediatric Asthma
Acronym: CLASSE
Status: Withdrawn | Type: Observational
Why Stopped: The study never started
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180357
Record Dates: First submitted 2018-11-02; First posted 2018-12-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-11

CONDITIONS: Severe Asthma
Keywords: Severe asthma in children; Type 2 innate lymphoid cells (ILC2); bronchial mucosa; bronchoalveolar lavages
MeSH Terms: conditions — Asthma | interventions — Biopsy; Blood Specimen Collection; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthmatic children: Severe uncontrolled asthma is defined by the need to maintain a treatment with high doses of inhaled corticosteroids and a long-acting bronchodilator (B2LDA) and/or an anti-leukotriene
  Interventions: Biological: Biopsy; Biological: Blood collection; Biological: Bronchoalveolar lavage
- Controls: Non-asthmatic children, paired in age, requiring bronchial endoscopy with BAL and bronchial mucosa biopsy.
  Interventions: Biological: Biopsy; Biological: Blood collection; Biological: Bronchoalveolar lavage

INTERVENTIONS:
Biological: Biopsy — Mucosal biopsies under general anesthesia of the segmental bronchi of the right or left lower lobe
Biological: Blood collection — Blood collection (+15mL/ current care)
Biological: Bronchoalveolar lavage — Bronchoalveolar lavage fluid (3mL/Kg)

SUMMARY:
The main objectives of this study are to show that the number of type 2 innate lymphoid cells (ILC2) of the bronchial mucosa and in bronchoalveolar lavages (BAL) are higher in asthmatic children than in non-asthmatics, that the number of ILC2 of the bronchial mucosa and in BAL correlate with the number of bronchial and BAL eosinophils, and to determine whether there is a correlation between plasma and bronchial and BAL ILC2.

DETAILED DESCRIPTION:
Severe asthma of the child is characterized by chronic eosinophilic infiltration of the bronchial mucosa associated with bronchial remodeling.

The mechanisms responsible for these phenomena are still misunderstood. Animal models suggest that type 2 innate lymphoid cells (ILC2) may be responsible for inflammation and bronchial remodeling in asthma. In mice, ILC2 stimulated by the pulmonary epithelium by viral aggression or allergenic exposure release cytokines of the TH2 type such as IL-5 and IL-13 and amphiregulin, involved in the recruitment and differentiation of eosinophils, bronchoconstriction, mucus secretion and the restoration of epithelial integrity.

In humans, ILC2 would be more abundant in the bronchoalveolar lavage (BAL) and peripheral blood of asthmatic patients compared to control subjects. However, the presence of ILC2 in the bronchial mucosa of asthmatic patients has never been identified.

The hypothesis tested is that ILC2 are more abundant in bronchial mucosa, BAL, and blood in children with severe asthma than in non-asthmatics. The results of this study would improve the knowledge of the mechanisms responsible for bronchial inflammation in asthma, consider therapies to prevent its development and modify the natural history of the disease.

The main objectives of this study are to show that the number of ILC2 in bronchial mucosa and BAL is higher in asthmatic children than in non-asthmatics, that the number of ILC2 in the bronchial mucosa and BAL is correlated with the number of eosinophils in bronchial mucosa and BAL, to determine whether the number of ILC2 in lungs correlate with asthma symptoms, and to determine whether there is a correlation between plasma and bronchial ILC2.

Bronchoscopy with BAL and bronchial mucosal biopsies will be performed in 20 children with severe asthma and 20 control subjects in the department of pediatric pulmonology and allergy of Necker Hospital.

ILC2 will be identified in the BAL, in the bronchial mucosa and peripheral blood by flow cytometry. The median values of the number of ILC2 will be compared between asthmatic and non-asthmatic patients by the Mann-Whitney non-parametric test. The correlations will be established by the Spearman rank test. A value of p < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

Controls :

* Minors aged 6 to 18 matched in age with severe asthmatic children
* Non-asthmatic children hospitalized in the department of pediatric pulmonology and allergy in Necker Hospital
* To undergo bronchial endoscopy with bronchoalveolar lavage, biopsy and blood collection

Severe asthmatic children :

* Minors aged 6 to 18
* Children hospitalized in the department of pediatric pulmonology and allergy in Necker Hospital
* To undergo bronchial endoscopy with bronchoalveolar lavage, biopsy and blood collection
* Severe uncontrolled asthma is defined by the need to maintain a treatment with high doses of inhaled corticosteroids and a long-acting bronchodilator (B2LDA) and/or an anti-leukotriene

Exclusion Criteria:

* Children with an immune deficiency, will be excluded

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minors hospitalized in the department of pediatric pulmonology and allergy of Necker Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Number of type 2 innate lymphoid cells | Day 0
  Type 2 innate lymphoid cells

SECONDARY OUTCOMES:
Number of Eosinophils | Day 0
  Eosinophils
Airway remodeling: reticular basement membrane thickness | Day 0
  Reticular basement membrane thickness will be expressed in µm.
Airway remodeling: airway smooth muscle area | Day 0
  The percentage of the submucosa occupied by airway smooth muscle will be determined on hematoxylin-eosin-stained and anti-airway smooth muscle antibody treated sections, respectively. The bundles of airway smooth muscle will be enclosed by a line and the area they occupied will be calculated by image analysis. The airway smooth muscle area will be expressed as the percentage of surface of the submucosa occupied by airway smooth muscle.
Airway remodeling: epithelial integrity | Day 0
  Epithelial integrity will be defined as the percentage of the total length of epithelium that will be intact.
Airway remodeling: vessel number | Day 0
  The number of vessels stained with anti-CD31 mAb will be determined from at least one grid (0.1 mm2) per biopsy, and reported as the median number of positive sections per 0.1 mm2.
Airway remodeling: mucus gland area | Day 0
  The percentage of the submucosa occupied by mucus gland will be determined on hematoxylin-eosin-stained and anti-airway smooth muscle antibody treated sections, respectively. The mucus glands will be enclosed by a line and the area occupied will be calculated by image analysis. The mucus gland area will be expressed as the percentage of surface of the submucosa occupied by mucus gland.
Airway inflammation: bronchoalveolar lavage (BAL) | Day 0
  BAL fluid will be assed for inflammation
  * The number of eosinophils will be assessed and expressed percentage of total cells in BAL
  * The number of neutrophils will be assessed and expressed percentage of total cells in BAL
  * The number of macrophages will be assessed and expressed percentage of total cells in BAL
  * The number of basophils will be assessed and expressed percentage of total cells in BAL
  * The number of mast cells will be assessed and expressed percentage of total cells in BAL
  * The number of innate lymphoid cells will be assessed and expressed percentage of total cells in BAL
  * The number of mucosal associated invariant T (MAIT) cells will be assessed and expressed percentage of total cells in BAL
  * The number of invariant natural killer T cells will be assessed and expressed percentage of total cells in BAL
  * The number of gammadelta T cells will be assessed and expressed percentage of total cells in BAL
Airway inflammation: bronchial mucosa | Day 0
  Bronchial sections will be stained with May-Grunwald-Giemsa.The number of inflammatory cells will be assessed in the submucosa and expressed as the number of cells per square millimeters of submucosal area.
  * The number of eosinophils will be assessed and expressed per square millimeters of submucosal area
  * The number of neutrophils in the submucosa will be assessed and expressed per square millimeters of submucosal area
  * The number of mast cells (c-kit positive cells) in the submucosa will be assessed and expressed per square millimeters of submucosal area
  * The number of IgE stained with anti-IgE Ab in the submucosa and the epithelium will be assessed and expressed per square millimeters of submucosal area
  * The expression of cytokines in the mucosa will be assessed by multiplex
Inflammation in blood | Day 0
  * The number of eosinophils will be assessed and expressed percentage of total cells in blood
  * The number of neutrophils will be assessed and expressed percentage of total cells in blood
  * The number of basophils will be assessed and expressed percentage of total cells in blood
  * The number of lymphocytes will be assessed and expressed percentage of total cells in blood
  * The number of innate lymphoid cells will be assessed and expressed percentage of total cells in blood
  * The number of mucosal associated invariant T (MAIT) cells will be assessed and expressed percentage of total cells and T cells in blood
  * The number of invariant natural killer T cells will be assessed and expressed percentage of total cells and T cells in blood
  * The number of gammadelta T cells will be assessed and expressed percentage of total cells and T cells in blood
  * The expression of cytokine will be assessed using multiplex analysis
Metabolomic signature | Day 0
  Non-targeted metabolomics analysis will be performed on plasma. Metabolic profiles will be obtained using two complementary LC-MS methods, to identify metabolites discriminating different patients.
Microbiota analysis | Day 0
  Microbiota analysis will be performed on BAL using PCR ARN 16S.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lezmi, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No